CLINICAL TRIAL: NCT04159766
Title: A Phase 2a Dose-Finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NLY01, a PEGylated Exenatide, When Administered as a Single Dose in Subjects With Type 2 Diabetes
Brief Title: A Study With NLY01 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuraly, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NLY01-D1
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Type2 Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- NLY01 (2.5 mg) (Active Comparator)
  Interventions: Drug: NLY01
- NLY01 (5.0 mg) (Active Comparator)
  Interventions: Drug: NLY01
- NLY01 (10 mg) (Active Comparator)
  Interventions: Drug: NLY01
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NLY01 — NLY01, a PEGylated form of the anti-diabetic peptide exenatide
  Arms: NLY01 (10 mg); NLY01 (2.5 mg); NLY01 (5.0 mg)
Drug: Placebo — normal saline
  Arms: Placebo

SUMMARY:
This is a Phase 2a study designed to assess the effect of NLY01 in patients with type 2 diabetes. Patients will be monitored for safety, pharmacokinetics, and pharmacodynamic effects on glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject with type 2 diabetes for at least one year
* Willing to continue treatment with metformin at the same dose and frequency until and (if applicable) to pause any treatment with a second oral antidiabetic
* Body Mass Index (BMI) 22.0 to 35.0 kg/m^2,

Exclusion Criteria:

* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
* Any history or presence of clinically relevant comorbidity (with the exception of conditions associated with diabetes mellitus), that may place the subject at increased risk as determined by the investigator
* Any prior exposure to an exenatide-based product (BYETTA and BYDUREON)
* History of gastroparesis
* History of severe hypoglycemia in the past 6 months
* If female, pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events | 35 days
Number of Incidences of Adverse Events | 35 days
Plasma glucose | 24 hours
  Change of fasting glucose profiles
Change in serum insulin | 24 hours
  Change in 24 hour serum insulin
Change in plasma glucagon | 24 hours
  Change in 24 hour plasma glucagon concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Dan Lee, Study Director — Neuraly, Inc.
Locations (2):
- Germany (2):
  - Profil Institute fur Stoffwechselforschung GmbH, Neuss
  - Profil Institute, Neuss